CLINICAL TRIAL: NCT00479167
Title: A Phase II Trial of Combined Weekly Bortezomib and Tositumomab I-131 in Patients With Relapsed or Refractory Follicular Non-Hodg
Brief Title: A Phase II Trial of Combined Weekly Bortezomib and Tositumomab I-131 in Patients With Relapsed or Refractory Follicular Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual and interest in study
Sponsor: Rush University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYM 2005-01
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Follicular Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Follicular Non-Hodgkin's Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma | interventions — Bortezomib; tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib and Tositumomab I-131 (Experimental)
  Interventions: Drug: Bortezomib and Tositumomab I-131

INTERVENTIONS:
Drug: Bortezomib and Tositumomab I-131

SUMMARY:
The purpose of this study is to determine what dose of bortezomib in combination with tositumomab I-131 is tolerable whether bortezomib and Tositumomab I-131 are effective in the treatment of relapsed or refractory non-hodgkin's lymphoma (NHL). Both agents are effective in treating relapsed and refractory NHL. Administer of the agents together may sensitize the cells to the radiation from Tositumomab I-131.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated or relapsed follicular lymphoma. One prior therapy required.
* Bi-dimensionally measurable disease with at least one lesion measuring > 2.0 X 2.0cm by CT scan or evaluable disease.
* CD20+ at time of diagnosis or subsequently.
* Platelet count > 100,000/uL, ANC > 1000/uL.
* Transaminases less than two-fold normal range.
* Adequate renal function defined as <1.5 X upper limit of normal
* HAMA negative
* ECOG performance status 0, 1, 2.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Negative Hepatitis profile screening

Exclusion Criteria:

* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to boron or mannitol.
* Greater than 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens
* Hypocellular bone marrow (≤15% cellularity or marked reduction in bone marrow precursors).
* Prior myeloablative therapy.
* History of failed stem cell collection.
* Prior radiotherapy to fields encompassing more than 25% of the blood-forming marrow.
* Prior chemotherapy, biologic therapy, radiation therapy or steroid therapy for NHL within three weeks prior to screening procedures. Six weeks for nitrosureas. Subjects receiving low doses of steroids for non-neoplastic indications may enter the study ("low dose steroids" is defined as ≤10 mg of prednisone or equivalent per day).
* Prior Radioimmunotherapy or bortezomib.
* Prior malignancy other than lymphoma, except for adequately treated basal cell or squamous cell skin cancer, in situ uterine cervical cancer, or other cancer for which the subject has been disease-free for five years.
* Evidence of active infection requiring intravenous antibiotics at the time of study enrollment.
* Known HIV infection.
* Known brain or leptomeningeal metastases.
* Active obstructive hydronephrosis.
* Known Type I hypersensitivity or anaphylactic reactions to murine proteins or any component of the Iodine I 131 tositumomab therapeutic regimen.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Gregory, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD, Maas J, Pien CS, Prakash S, Elliott PJ. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res. 1999 Jun 1;59(11):2615-22. PMID 10363983
- [Background] Cusack JC Jr, Liu R, Houston M, Abendroth K, Elliott PJ, Adams J, Baldwin AS Jr. Enhanced chemosensitivity to CPT-11 with proteasome inhibitor PS-341: implications for systemic nuclear factor-kappaB inhibition. Cancer Res. 2001 May 1;61(9):3535-40. PMID 11325813
- [Background] Fossella FV, DeVore R, Kerr RN, Crawford J, Natale RR, Dunphy F, Kalman L, Miller V, Lee JS, Moore M, Gandara D, Karp D, Vokes E, Kris M, Kim Y, Gamza F, Hammershaimb L. Randomized phase III trial of docetaxel versus vinorelbine or ifosfamide in patients with advanced non-small-cell lung cancer previously treated with platinum-containing chemotherapy regimens. The TAX 320 Non-Small Cell Lung Cancer Study Group. J Clin Oncol. 2000 Jun;18(12):2354-62. doi: 10.1200/JCO.2000.18.12.2354. PMID 10856094
- [Background] Hideshima T, Richardson P, Chauhan D, Palombella VJ, Elliott PJ, Adams J, Anderson KC. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res. 2001 Apr 1;61(7):3071-6. PMID 11306489
- [Background] Jagannath S, Barlogie B, Berenson J, Siegel D, Irwin D, Richardson PG, Niesvizky R, Alexanian R, Limentani SA, Alsina M, Adams J, Kauffman M, Esseltine DL, Schenkein DP, Anderson KC. A phase 2 study of two doses of bortezomib in relapsed or refractory myeloma. Br J Haematol. 2004 Oct;127(2):165-72. doi: 10.1111/j.1365-2141.2004.05188.x. PMID 15461622
- [Background] LeBlanc R, Catley LP, Hideshima T, Lentzsch S, Mitsiades CS, Mitsiades N, Neuberg D, Goloubeva O, Pien CS, Adams J, Gupta D, Richardson PG, Munshi NC, Anderson KC. Proteasome inhibitor PS-341 inhibits human myeloma cell growth in vivo and prolongs survival in a murine model. Cancer Res. 2002 Sep 1;62(17):4996-5000. PMID 12208752
- [Background] Lightcap ES, McCormack TA, Pien CS, Chau V, Adams J, Elliott PJ. Proteasome inhibition measurements: clinical application. Clin Chem. 2000 May;46(5):673-83. PMID 10794750
- [Background] Orlowski RZ, Stinchcombe TE, Mitchell BS, Shea TC, Baldwin AS, Stahl S, Adams J, Esseltine DL, Elliott PJ, Pien CS, Guerciolini R, Anderson JK, Depcik-Smith ND, Bhagat R, Lehman MJ, Novick SC, O'Connor OA, Soignet SL. Phase I trial of the proteasome inhibitor PS-341 in patients with refractory hematologic malignancies. J Clin Oncol. 2002 Nov 15;20(22):4420-7. doi: 10.1200/JCO.2002.01.133. PMID 12431963
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Teicher BA, Ara G, Herbst R, Palombella VJ, Adams J. The proteasome inhibitor PS-341 in cancer therapy. Clin Cancer Res. 1999 Sep;5(9):2638-45. PMID 10499643
- [Background] Press OW, Appelbaum F, Ledbetter JA, Martin PJ, Zarling J, Kidd P, Thomas ED. Monoclonal antibody 1F5 (anti-CD20) serotherapy of human B cell lymphomas. Blood. 1987 Feb;69(2):584-91. PMID 3492224
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] Young RC, Longo DL, Glatstein E, Ihde DC, Jaffe ES, DeVita VT Jr. The treatment of indolent lymphomas: watchful waiting v aggressive combined modality treatment. Semin Hematol. 1988 Apr;25(2 Suppl 2):11-6. PMID 2456618
- [Background] Horning SJ. Natural history of and therapy for the indolent non-Hodgkin's lymphomas. Semin Oncol. 1993 Oct;20(5 Suppl 5):75-88. No abstract available. PMID 8211209
- [Background] Yuen AR, Kamel OW, Halpern J, Horning SJ. Long-term survival after histologic transformation of low-grade follicular lymphoma. J Clin Oncol. 1995 Jul;13(7):1726-33. doi: 10.1200/JCO.1995.13.7.1726. PMID 7602362
- [Background] Gallagher CJ, Gregory WM, Jones AE, Stansfeld AG, Richards MA, Dhaliwal HS, Malpas JS, Lister TA. Follicular lymphoma: prognostic factors for response and survival. J Clin Oncol. 1986 Oct;4(10):1470-80. doi: 10.1200/JCO.1986.4.10.1470. PMID 3531422
- [Background] McKelvey EM, Gottlieb JA, Wilson HE, Haut A, Talley RW, Stephens R, Lane M, Gamble JF, Jones SE, Grozea PN, Gutterman J, Coltman C, Moon TE. Hydroxyldaunomycin (Adriamycin) combination chemotherapy in malignant lymphoma. Cancer. 1976 Oct;38(4):1484-93. doi: 10.1002/1097-0142(197610)38:43.0.co;2-i. PMID 791473
- [Background] Johnson PW, Rohatiner AZ, Whelan JS, Price CG, Love S, Lim J, Matthews J, Norton AJ, Amess JA, Lister TA. Patterns of survival in patients with recurrent follicular lymphoma: a 20-year study from a single center. J Clin Oncol. 1995 Jan;13(1):140-7. doi: 10.1200/JCO.1995.13.1.140. PMID 7799014
- [Background] White CA, Weaver RL, Grillo-Lopez AJ. Antibody-targeted immunotherapy for treatment of malignancy. Annu Rev Med. 2001;52:125-45. doi: 10.1146/annurev.med.52.1.125. PMID 11160771
- [Background] Demidem A, Lam T, Alas S, Hariharan K, Hanna N, Bonavida B. Chimeric anti-CD20 (IDEC-C2B8) monoclonal antibody sensitizes a B cell lymphoma cell line to cell killing by cytotoxic drugs. Cancer Biother Radiopharm. 1997 Jun;12(3):177-86. doi: 10.1089/cbr.1997.12.177. PMID 10851464
- [Background] Press OW, Rasey J. Principles of radioimmunotherapy for hematologists and oncologists. Semin Oncol. 2000 Dec;27(6 Suppl 12):62-73. PMID 11226002
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Background] Kaminski MS, Zasadny KR, Francis IR, Fenner MC, Ross CW, Milik AW, Estes J, Tuck M, Regan D, Fisher S, Glenn SD, Wahl RL. Iodine-131-anti-B1 radioimmunotherapy for B-cell lymphoma. J Clin Oncol. 1996 Jul;14(7):1974-81. doi: 10.1200/JCO.1996.14.7.1974. PMID 8683227
- [Background] Shan D, Ledbetter JA, Press OW. Apoptosis of malignant human B cells by ligation of CD20 with monoclonal antibodies. Blood. 1998 Mar 1;91(5):1644-52. PMID 9473230
- [Background] Buchsbaum DJ, Wahl RL, Normolle DP, Kaminski MS. Therapy with unlabeled and 131I-labeled pan-B-cell monoclonal antibodies in nude mice bearing Raji Burkitt's lymphoma xenografts. Cancer Res. 1992 Dec 1;52(23):6476-81. PMID 1423295
- [Background] Davis TA, Grillo-Lopez AJ, White CA, McLaughlin P, Czuczman MS, Link BK, Maloney DG, Weaver RL, Rosenberg J, Levy R. Rituximab anti-CD20 monoclonal antibody therapy in non-Hodgkin's lymphoma: safety and efficacy of re-treatment. J Clin Oncol. 2000 Sep;18(17):3135-43. doi: 10.1200/JCO.2000.18.17.3135. PMID 10963642
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib in Combination With Tositumomab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: only subject withdrew
Arm/Group | Bortezomib in Combination With Tositumomab
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Study is to Determine the Maximum Tolerated Dose (up to 1.6 mg/m2) of Bortezomib Combined With Tositumomab and Iodine I 131 Tositumomab
Time Frame: Study terminated.
Population: Subject withdrew
Groups:
- Bortezomib Combined With Tositumomab and Iodine I 131 Tositumomab: Bortezomib Combined With Tositumomab and Iodine I 131 Tositumomab
Arm/Group | Bortezomib Combined With Tositumomab and Iodine I 131 Tositumomab
Number analyzed (Participants) | 0

2. Secondary Outcome: To Further Explore the Toxicity and Efficacy of Bortezomib Combined With Tositumomab and Iodine I 131 Tositumomab and Assess the Tolerability of Bortezomib After Tositumomab
Time Frame: Study Terminated.
Population: Subject withdrew
Groups:
- Bortezomib and Tositumomab I-131: Bortezomib and Tositumomab I-131
Arm/Group | Bortezomib and Tositumomab I-131
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Bortezomib in Combination With Tositumomab: Bortezomib in combination with tositumomab
Arm/Group | Bortezomib in Combination With Tositumomab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Only 1 patient was on study and withdrew after 1 cycle. There was lack of interest in the study. The PI is now retiring.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes